CLINICAL TRIAL: NCT03276104
Title: Late In-the-bag intraOcular Lens dislocatioN Surgery: A Randomized Clinical Trial (LION Trial)
Brief Title: Late In-the-bag intraOcular Lens dislocatioN Surgery
Acronym: LION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Marius Dalby, Principal Investigator, M.D., PhD Candidate, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/5506
Record Dates: First submitted 2017-08-31; First posted 2017-09-08 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Intraocular Lens Dislocation
Keywords: IOL dislocation; Cataract; Cataract surgery; Scleral suturing; Verisyse; Iris-claw; Late in-the-bag IOL dislocation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Masking of research optometrists to group affiliation at the postoperative examinations will be endeavored. A physician will perform slit lamp examinations at the postoperative visits, hence he/she cannot be masked, nor can the surgeon. The investigator will be masked during the image analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL repositioning group (Active Comparator)
  Interventions: Procedure: IOL repositioning
- IOL exchange group (Active Comparator)
  Interventions: Procedure: IOL exchange

INTERVENTIONS:
Procedure: IOL repositioning — Intraocular lens repositioning by scleral suturing
  Arms: IOL repositioning group
Procedure: IOL exchange — Intraocular lens exchange with retropupillary iris-claw lens
  Arms: IOL exchange group

SUMMARY:
Overall aim of the study is to compare the safety and efficacy of two different surgical methods to treat Late In-the-bag intraocular lens dislocation.

DETAILED DESCRIPTION:
Cataract is a condition of unclear lens that cause poor vision. The only treatment is surgery where the blurred biological lens is replaced with an artificial clear lens (IOL). Most people who operate achieve full vision. Nevertheless, serious complications may occasionally occur, and one of these is dislocation of the entire complex with IOL and lens capsule. This requires surgical treatment.

In this study the investigators want to compare two different surgical methods used in late dislocation of IOL inside the capsule after cataract surgery. Patients will be randomly affiliated to either the suturing of existing IOL / capsule complex, or lens exchange to an IOL fixed to the iris.

The focus of the trial will be especially on complications and other eye changes in the early stages of surgery. Today, little data is available on these topics, and the investigators believe that new knowledge can bring us closer to a response to preferred operating techniques and an optimal drug drop regime for the patient group.

ELIGIBILITY:
Inclusion Criteria:

* IOL inside the capsule ("in-the-bag")
* Late dislocation (more than 6 months after cataract surgery)
* IOL visible in the pupillary area in the supine position and hence possible to perform surgery with an anterior approach
* Eligibility for both operation methods
* Ability to cooperate fairly well during the examinations
* Willing to participate in the study, e.g. willingness to participate at all control visits

Exclusion Criteria:

* IOL designs that cannot be repositioned with a suture loop, such as plate-haptic IOLs without holes in the peripheral part
* Eyes with especially thin sclera
* Active uveitis or pronounced iris pathology
* Eyes with previously performed Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK)
* Totally dislocated IOL into the posterior segment of the eye requiring pars plana vitrectomy
* Eyes that prior to cataract extraction had a subluxated lens in need of surgery with a Cionni capsular tension ring (e.g. patients with Marfan syndrome and ectopia lentis)
* Cases requiring a change in refraction. Risk of severe anisometropia
* Patients unable to lie in supine position for surgery in local anesthesia, e.g. severe chronic obstructive pulmonary disease and severe heart failure
* Patients using anticoagulants that cannot be discontinued

For patients with dislocated IOLs in both eyes during the study period, only the first operated eye will be included. Patients without prospects of improvement in vision will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-09 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Inflammation in the anterior chamber after surgery | The first weeks after surgery
  Measured with a Laser Flare Meter
Changes in macular thickness and occurrence of Cystoid macular edema | The first months after surgery, and long term changes months up to two years after surgery
  Evaluated with Optical Coherence Tomography
Intraocular pressure changes | Early changes in the first weeks after surgery, and long term changes months up to two years after surgery
  Measured with Goldmann Applanation Tonometry and iCare, both measured in mmhg

SECONDARY OUTCOMES:
Best Corrected Visual acuity (BCVA) | Short term (the first weeks and up to 6 months) and long term (up to two years)
  Measured in LogMar
Best Corrected Visual acuity (BCVA) | Short term (the first weeks and up to 6 months) and long term (up to two years)
  Measured in Snellen
Glare | Medium term (6 months)
  Measured by straylight meter
Glare | Medium term (6 months)
  Measured by subjective presence of glare
Endothelial cells | Short term (2 weeks) and long term (6months and 2 years)
  Measured by Non-contact corneal confocal microscopy
Intra- and postoperative complications | Short term and long term (first post operative day, the first weeks and months, and up to two years)
  All relevant complications
IOL tilt | 6 months and 2 years
  Measured with anterior segment Ultra Sound
IOL tilt | 6 months and 2 years
  Measured with Anterior segment optical coherence tomography
Refractive outcomes - subjective refraction measured with a phoropter | Short term - meaning 2 weeks to 6 months. Long term - meaning up to two years
  To compare the refractive outcomes (short and long-term)
Refractive outcomes - subjective refraction measured with a phoropter | Short term - meaning 2 weeks to 6 months. Long term - meaning up to two years
  To determine whether suture placement for IOL repositioning affects the refractive outcome
Astigmatism | Short term - meaning 2 weeks to 6 months. Long term - meaning up to two years
  To compare astigmatism measured by keratometry
Astigmatism | Short term - meaning 2 weeks to 6 months. Long term - meaning up to two years
  To compare astigmatism measured by subjective refraction measured with phoropter

CONTACTS AND LOCATIONS:
Overall Officials: Liv Drolsum, Prof. M.D. PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No